CLINICAL TRIAL: NCT05904210
Title: Retrospective Experience Assessing the Real-World Utilization and Effectiveness of SEVENFACT® [Coagulation Factor VIIa (Recombinant) - Jncw] in the USA
Brief Title: Retrospective Experience Assessing the Real-World Utilization and Effectiveness of SEVENFACT®
Status: Completed | Type: Observational
Sponsor: Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Responsible Party: Sponsor
Other Study IDs: F7TG2204
Record Dates: First submitted 2023-05-16; First posted 2023-06-15 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Hemophilia
Keywords: inhibitors; eptacog beta; recombinant factor 7; real-world evidence
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated by SEVENFACT®: Patients that initiated treatment with SEVENFACT® in real-world clinical care in the USA will be eligible.
  Data from eligible patients' medical charts, bleeding diaries, and medication logs will be extracted from the time of initiation of SEVENFACT® treatment and for each bleeding episode and surgery or invasive procedure requiring treatment with SEVENFACT® or for prophylaxis, up until the data collection at the investigational site.
  Interventions: Drug: SEVENFACT®

INTERVENTIONS:
Drug: SEVENFACT® — Coagulation Factor VIIa (Recombinant)

SUMMARY:
Retrospective Experience Assessing the Real-World Utilization and Effectiveness of SEVENFACT® [coagulation factor VIIa (recombinant)-jncw] in the USA.

The current study will provide a unique opportunity to describe the profile of the early patients selected for treatment with SEVENFACT® and to assess the real-world utilization (effectiveness, safety, tolerability, and modalities of treatment) of SEVENFACT®.

DETAILED DESCRIPTION:
Parameters collected will include patient socio-demographics, medical history / comorbidities, bleeding disorder history, physical examination, vital signs, prior and concomitant bleeding disorder treatments, bleeding episode / surgery or invasive procedure / prophylaxis details, information on SEVENFACTâ treatment modalities, retrospective investigator rating of SEVENFACTâ effectiveness using the Clinical Global Impression Efficacy Index (CGI-E) and time for bleed control, Adverse Drug Experiences (ADEs) temporally associated with SEVENFACTâ administration, special situations that occurred during SEVENFACTâ administration, whether or not associated with ADE, laboratory testing for activation of the coagulation system or thrombosis, physical examination, and vital signs.

ELIGIBILITY:
Inclusion Criteria:

1. Patient received SEVENFACT® before study initiation.
2. If collection of a written informed consent is required for an investigational site (see Section 5.1 General Informed Consent), patient has read, understood, and documented written informed consent/assent.

Exclusion Criteria:

Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Full Analysis Set (FAS) defined as all patients that received at least one dose of SEVENFACT®. Missing data will not be imputed, and all analyses will be based on observed data only.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-05-09 (Actual); Study Completion 2024-05-09 (Actual)

PRIMARY OUTCOMES:
SEVENFACT® effectiveness | For all events which took place from Jan 1st, 2021 up to site opening in 2023
  SEVENFACT® effectiveness will be evaluated based on the retrospective rating by the investigator using the Clinical Global Impression Efficacy Index (CGI-E) for each 'event' (bleeding episode, surgery or invasive procedure, or prophylaxis). Specifically, the proportion of patients receiving efficient treatment based on CGI-E will be estimated.

SECONDARY OUTCOMES:
Patient profile analysis | For all events which took place from Jan 1st, 2021 up to site opening in 2023
  The patient profile of patients treated with SEVENFACT® will be evaluated based on the patient's socio-demography, medical history, potential comorbidities, physical examination, current medications, and bleeding disorder history

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Luskin Orthopaedic Institute for Children, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Children's healthcare of Atlanta, Atlanta, Georgia
  - Mayo Clinic, Rochester, Minnesota
  - SUNY Upstate Medical University, Pediatric Hematology/Oncology, Syracuse, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The Gulf States Hemophilia & Thrombophilia Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang M, Lawrence JB, Quon DV, Ducore J, Simpson ML, Boggio LN, Mitchell IS, Yuan G, Alexander WA, Schved JF. PERSEPT 1: a phase 3 trial of activated eptacog beta for on-demand treatment of haemophilia inhibitor-related bleeding. Haemophilia. 2017 Nov;23(6):832-843. doi: 10.1111/hae.13301. Epub 2017 Aug 3. PMID 28776894